CLINICAL TRIAL: NCT02113670
Title: Changes in Abdominal Leak Point Pressures in Women Stress Urinary Incontinence Following Intravesical Air Instillation During Urodynamic Study
Brief Title: Changes in ALPP in Women With SUI Following Air Instillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Collaborators: The Trendlines Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TrendLinesSUI
Record Dates: First submitted 2014-03-28; First posted 2014-04-14 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; abdominal leak point pressure; urodynamic study
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SUI 1 (Experimental): Patients will perform urodynamic study before and after instillation of 50 ml of air
  Interventions: Other: SUI 1

INTERVENTIONS:
Other: SUI 1 — instillation of 50ml of air into the urinary bladder before the urodynamic test
  Other Names: 50ml of air instillation into the bladder

SUMMARY:
More than 11 million women in the United States suffer from stress urinary incontinence (SUI), the involuntary leakage of urine during everyday activities that put temporary stress on the abdomen and bladder, such as laughing, coughing, and walking. For women with SUI, this pressure often causes urine to leak involuntarily. SUI affects women of all ages including young mothers, pre-menopausal women, and seniors, and can result in significant emotional distress. Current solutions for SUI include disposable pads, behavioral treatment (pelvic floor physical therapy) and surgical intervention. Patients with SUI who failed conservative treatment and wish to be further treated by a surgery may require further work-up by urodynamic study in which abdominal leak point pressures (ALPP) defined and reflect the severity of SUI.

There is continuous need to develop less invasive treatments for SUI that could minimize the use of pads, could be an alternative to painful, costly surgical procedure. The Trendlines Group lab solution is a non-surgical alternative in the treatment of SUI. The concept of the future treatment solution is based on simple physics: injecting a small amount of air into the urinary bladder, which eliminates or greatly reduces involuntary urinary leakage. The air bubble acts as a "shock absorber" to reduce the temporary pressure increase in the bladder that causes urinary leakage. The concept for the new treatment has been tested in a lab environment using lab jig tests and pig urinary system (bladder and urethra). The lab tests showed significant improvement in the bladder pressure when the treatment was implemented by suspending the stress pressure to a level that will not cause urine leakage.

DETAILED DESCRIPTION:
More than 11 million women in the United States suffer from stress urinary incontinence (SUI), the involuntary leakage of urine during everyday activities that put temporary stress on the abdomen and bladder, such as laughing, coughing, and walking. For women with SUI, this pressure often causes urine to leak involuntarily. SUI affects women of all ages including young mothers, pre-menopausal women, and seniors, and can result in significant emotional distress. Current solutions for SUI include disposable pads, behavioral treatment (pelvic floor physical therapy) and surgical intervention. Patients with SUI who failed conservative treatment and wish to be further treated by a surgery may require further work-up by urodynamic study in which abdominal leak point pressures (ALPP) defined and reflect the severity of SUI.

There is continuous need to develop less invasive treatments for SUI that could minimize the use of pads, could be an alternative to painful, costly surgical procedure. The Trendlines Group lab solution is a non-surgical alternative in the treatment of SUI. The concept of the future treatment solution is based on simple physics: injecting a small amount of air into the urinary bladder, which eliminates or greatly reduces involuntary urinary leakage. The air bubble acts as a "shock absorber" to reduce the temporary pressure increase in the bladder that causes urinary leakage. The concept for the new treatment has been tested in a lab environment using lab jig tests and pig urinary system (bladder and urethra). The lab tests showed significant improvement in the bladder pressure when the treatment was implemented by suspending the stress pressure to a level that will not cause urine leakage.

Following positive results of this proof of concept study we could plan further innovative device to treat SUI in women.

ELIGIBILITY:
Inclusion Criteria:

1. Women
2. Age >18 years old
3. SUI: pure or stress predominant mixed urinary incontinence.
4. Failure of conservative treatment who desires surgical procedure for SUI.
5. Signed informed consent for the trial and urodynamic study.
6. Negative urine culture.

Exclusion Criteria:

1. Neurogenic SUI
2. Unable or unwilling to sign informed consent for the trial and urodynamic study.
3. Patient who does not will a surgery for SUI
4. Prior pelvic or lower abdominal malignancies
5. Prior pelvic radiation or surgery except anterior/posterior colporrhaphy or hysterectomy (with or without oophorectomy) for benign disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
change in abdominal leak point pressure | 1 day
  to verify the concept of a possible future treatment in the clinical setup by checking physical effect of dumping pressure (decrease in ALLP) by inserting 50 ml of air into the bladder during the urodynamic study in patients with SUI.

SECONDARY OUTCOMES:
adverse events as a measure of safety and tolerability | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel